CLINICAL TRIAL: NCT06333639
Title: Implementing Virtual Reality in the Operating Room : Patient Satisfaction During Long Orthopaedic Surgery Under Locoregional Anaesthesia
Brief Title: Implementing Virtual Reality in the Operating Room
Acronym: IRVABO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24Chirortho01
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: General Surgery; Orthopedic Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- orthopaedic surgery (goup 1 control): 30 individuals installed according to the usual procedures for an orthopaedic surgery
  Interventions: Other: orthopaedic surgery
- orthopaedic surgery and fitted with a virtual reality headset (group 2 case): 30 individuals installed according to the usual procedures for an orthopaedic surgery and fitted with a virtual reality headset
  Interventions: Other: orthopaedic surgery and fitted with a virtual reality headset

INTERVENTIONS:
Other: orthopaedic surgery — usual procedures for an orthopaedic surgery
  Groups: orthopaedic surgery (goup 1 control)
Other: orthopaedic surgery and fitted with a virtual reality headset — usual procedures for an orthopaedic surgery and fitted with a virtual reality headset
  Groups: orthopaedic surgery and fitted with a virtual reality headset (group 2 case)

SUMMARY:
"Recently, virtual reality has become more accessible thanks to the use of smaller, more comfortable and easier-to-use devices. Its use in operating theatres is growing.

However, despite the clinical effectiveness of virtual reality in reducing pain and anxiety, there are very few feedback studies from patients on their experience of surgery and their satisfaction, especially in orthopaedics.

The aim of this study is to demonstrate the superiority, during long awake orthopaedic surgery, of equipping the patient with a virtual reality headset, on patient satisfaction, compared with the same surgery without a headset.

The visual support offered will be appropriate to the duration of the surgery, i.e. more than 1 hour."

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Patient admitted for total hip or knee replacement surgery.
* Patient undergoing anaesthetic management by loco-regional anaesthesia
* Affiliation to a French health insurance scheme or equivalent
* Patient who has given his non-opposition agreement

Exclusion Criteria:

* Patient with a neurological disorder (coma, dementia, confusion, photosensitive epilepsy)
* Patient with a severe psychiatric disorder
* Patients with severe deafness or visual impairment
* Language barrier
* Pregnant or breast-feeding women of childbearing age
* Refusal of patient involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients admitted for total hip or knee replacement surgery and whose anaesthetic management is by loco-regional anaesthesia
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
To demonstrate the superiority, during long awake orthopaedic surgery, of equipping the patient with a virtual reality headset, on patient satisfaction, compared with the same surgery without a headset. | Immediate post-operative
  Patient satisfaction with their surgical experience. This will be measured using a Likert scale, graduated from 0 to 10, with 0 being the minimum and 10 the maximum.

SECONDARY OUTCOMES:
1. To demonstrate the superiority, during long awake orthopaedic surgery, of equipping the patient with a virtual reality headset, on the doses of premedication, compared with the same surgeries without headset. | Immediate post-operative
  1. The number and doses of Midazolam (in mg) received in the two distinct groups will make it possible to evaluate the effectiveness of virtual reality from a pharmaceutical point of view. A difference in the use of pharmaceutical therapeutics of 20% less in patients with VR is expected to be significant. If the difference is less, the doses of premedication used in the two groups will be compared in order to assess the positive impact of VR.
Evaluate the Virtual Reality device in terms of comfort when wearing the headset, visual comfort and image and scenario quality, and auditory quality | Immediate post-operative
  2. VR evaluated using a Likert scale from 0 to as well as an open-ended questionnaire evaluating (isolation from noise pollution, possibility of communicating with nursing staff, quality of audio transmitted) : The comfort of wearing the helmet Visual comfort, image and scenario quality Hearing quality (isolation from noise pollution, ability to communicate with nursing staff, quality of audio transmitted)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NiICE, Nice, Alpes Maritimes, France